CLINICAL TRIAL: NCT00362479
Title: A Prospective, Multicenter, Open-Label Study to Evaluate the Safety and Efficacy of the 28-Day Oral Contraceptive DR-1021
Brief Title: Open-Label Study to Evaluate the Safety and Efficacy of a Low-Dose 28-Day Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DR-DSG-301
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Contraception
Keywords: pregnancy prevention; oral contraceptives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: DR-1021

INTERVENTIONS:
Drug: DR-1021 — 1 tablet daily

SUMMARY:
This is an open-label, single treatment study. All subjects will receive 6 months of oral contraceptive therapy with DR-1021. Study participants will receive physical and gynecological exams, including Pap smear. During the study, all participants will be required to complete a diary.

DETAILED DESCRIPTION:
The overall study duration for each patient will be approximately 8 months, which includes a screening period of approximately 4 weeks; a treatment period of approximately six months (six,28-day cycles); and a follow-up visit approximately 4 weeks after completion of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Not pregnant or breastfeeding
* Sexually active at risk of pregnancy

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy within the last 3 months
* Smoking > 10 cigarettes per day

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1347 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of pregnancy rates | Duration of study

SECONDARY OUTCOMES:
Adverse events reported by patients and investigators | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Medical Monitor, Principal Investigator — Duramed Research
Locations (79):
- United States (79):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Mobile, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Carmichael, California
  - Duramed Investigational Site, Irvine, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, San Ramon, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Lakewood, Colorado
  - Duramed Investigational Site, Wilmington, Delaware
  - Duramed Investigational Site, Washington D.C., District of Columbia
  - Duramed Investigational Site, Aventura, Florida
  - Duramed Investigational Site, Boynton Beach, Florida
  - Duramed Investigational Site, Brooksville, Florida
  - Duramed Investigational Site, Clearwater, Florida
  - Duramed Investigational Site, Coral Gables, Florida
  - Duramed Investigational Site, Fort Meyers, Florida
  - Duramed Investigational Site, Leesburg, Florida
  - Duramed Investigational Site, Longwood, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Pinellas Park, Florida
  - Duramed Investigational Site, Sarasota, Florida
  - Duramed Investigational Site, St. Petersburg, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Atlanta, Georgia
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Roswell, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Peoria, Illinois
  - Duramed Investigational Site, Shawnee Mission, Kansas
  - Duramed Investigational Site, Topeka, Kansas
  - Duramed Investigational Site, Lexington, Kentucky
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Mount Sterling, Kentucky
  - Duramed Investigational Site, Kansas City, Missouri
  - Duramed Investigational Site, Lincoln, Nebraska
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, New Brunswick, New Jersey
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Johnson City, New York
  - Duramed Investigational Site, Rochester, New York
  - Duramed Investigational Site, Charlotte, North Carolina
  - Duramed Investigational Site, Raleigh, North Carolina
  - Duramed Investigational Site, Wilmington, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Reading, Pennsylvania
  - Duramed Investigational Site, Cranston, Rhode Island
  - Duramed Investigational Site, Greer, South Carolina
  - Duramed Investigational Site, Mt. Pleasant, South Carolina
  - Duramed Investigational Site, Bristol, Tennessee
  - Duramed Investigational Site, Chattanooga, Tennessee
  - Duramed Investigational Site, Clarksville, Tennessee
  - Duramed Investigational Site, Germantown, Tennessee
  - Duramed Investigational Site, Knoxville, Tennessee
  - Duramed Investigational Site, Nashville, Tennessee
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Waco, Texas
  - Duramed Investigational Site, Magna, Utah
  - Duramed Investigational Site, Pleasant Grove, Utah
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Sandy City, Utah
  - Duramed Investigational Site, Arlington, Virginia
  - Duramed Investigational Site, Newport News, Virginia
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Richmond, Virginia
  - Duramed Investigational Site, Lakewood, Washington
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington